CLINICAL TRIAL: NCT00235040
Title: Evaluating Smart Forms and Quality Dashboards in an EHR: Effectiveness of the Acute Respiratory Infection Smart Form
Brief Title: Evaluating the Effectiveness of the Acute Respiratory Infection Smart Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Blackford Middleton, M.D., M.P.H, M.Sc., Partners Healthcare Systems, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HS015169-1; R01HS015169 (AHRQ)
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Respiratory Tract Infections
Keywords: Upper Respiratory Infections; Respiratory Tract Infections; Tree Number C01.539.739; Tree Number C08.730; Unique ID D012141
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Intervention
  Interventions: Behavioral: Smart Form
- 2 (No Intervention): Control
  Interventions: Behavioral: Smart Form

INTERVENTIONS:
Behavioral: Smart Form — Computer Decision Support System

SUMMARY:
To evaluate the effectiveness of the Acute Respiratory Infection Smart Form

DETAILED DESCRIPTION:
Specific Aim 1: To design and implement an integrated documentation-based clinical decision support and physician feedback system, provided in an electronic health record (EHR), to improve the management of patients with acute medical conditions.

Hypothesis 1: A documentation-based clinical decision support tool (CDSS) "smart form" physician feedback system, can be designed and implemented to facilitate documentation and physician order-entry, provide individualized, evidence-based recommendations for the management of patients acute respiratory infections (ARIs), and are usable by primary care physicians.

Specific Aim 2: To determine the effectiveness of documentation-based CDSS and physician feedback on documentation and the clinical management of patients respiratory tract infections.

Hypothesis 2A: A documentation-based CDSS "smart form" will increase the documentation of important clinical data in patients with ARI when compared to usual practice.

Hypothesis 2B: A documentation-based CDSS "smart form" will increase adherence with guidelines for the management of patients with ARI when compared to usual practice.

ELIGIBILITY:
Inclusion Criteria:

Acute Respiratory Infection visit

Exclusion Criteria:

Any patients who are not part of a panel of a participating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18257 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing rates | 9 months

SECONDARY OUTCOMES:
Appropriateness of antibiotic prescribing, re-visit rates, antibiotic costs, use of antibiotics, all-cause antibiotic use, quality of documentation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Blackford Middleton, MD, MPH, MSc, Principal Investigator — Partners Healthcare Systems Inc

REFERENCES:
- [Derived] Linder JA, Schnipper JL, Middleton B. Method of electronic health record documentation and quality of primary care. J Am Med Inform Assoc. 2012 Nov-Dec;19(6):1019-24. doi: 10.1136/amiajnl-2011-000788. Epub 2012 May 19. PMID 22610494